CLINICAL TRIAL: NCT02779738
Title: The Effect of Food on the Bioavailability of Merestinib in Healthy Subjects
Brief Title: A Study of Merestinib (LY2801653) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16439; I3O-MC-JSBH (Other: Eli Lilly and Company.)
Record Dates: First submitted 2016-05-19; First posted 2016-05-20 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
MeSH Terms: interventions — merestinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Merestinib Fasted (Experimental): Single dose of merestinib administered in fasted state in one of three periods
  Interventions: Drug: Merestinib
- Merestinib Standard Meal (Experimental): Single dose of merestinib administered with a standard meal in one of three periods
  Interventions: Drug: Merestinib
- Merestinib High-Fat Meal (Experimental): Single dose of merestinib administered with a high-fat meal in one of three periods
  Interventions: Drug: Merestinib

INTERVENTIONS:
Drug: Merestinib — Administered orally
  Other Names: LY2801653

SUMMARY:
The purpose of this study is to evaluate the effect of food on merestinib (standard meal and high-fat meal) compared to the fasted state. The study will also measure how much of the study drug gets into the blood stream and how long it takes the body to get rid of it. In addition, the tolerability of the study drug will be evaluated. Information about any side effects that may occur will also be collected. The study will last approximately 28 days. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy sterile male and female participants
* Body mass index (BMI) of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Are willing and able to eat the protocol specified high-fat breakfast

Exclusion Criteria:

* Have consumed grapefruits or grapefruit-containing products, Seville oranges or Seville orange juice, star fruit, star fruit juice, or star fruit-containing products, or commercial apple or orange juice within 14 days prior to first dosing
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have donated blood of more than 500 milliliters (mL) within the last month
* Cannot stop taking over-the-counter (OTC) or prescription medications that alter gastric pH, at least 14 days prior to first dosing
* Have previously completed or withdrawn from this study or any other study investigating merestinib, and have previously received the investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) for Merestinib for High-Fat Meal and Fasted State | Predose through 120 hours after administration of study drug
Pharmacokinetics: Maximum Concentration (Cmax) for Merestinib for Standard Meal and Fasted State | Predose through 120 hours after administration of study drug
Pharmacokinetics: Area Under The Concentration Curve AUC(0-∞) for Merestinib for High-Fat Meal and Fasted State | Predose through 120 hours after administration of study drug
Pharmacokinetics: Area Under The Concentration Curve AUC(0-∞) for Merestinib for Standard Meal and Fasted State | Predose through 120 hours after administration of study drug

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) for Metabolites (M1 and M2) for High-Fat Meal and Fasted State | Predose through 120 hours after administration of study drug
Pharmacokinetics: Maximum Concentration (Cmax) for Metabolites (M1 and M2) for Standard Meal and Fasted State | Predose through 120 hours after administration of study drug
Pharmacokinetics: Area Under the Concentration Curve AUC(0-∞) for Metabolites (M1 and M2) for High-Fat Meal and Fasted State | Predose through 120 hours after administration of study drug
Pharmacokinetics: Area Under the Concentration Curve AUC(0-∞) for Metabolites (M1 and M2) for Standard Meal and Fasted State | Predose through 120 hours after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States